CLINICAL TRIAL: NCT03860116
Title: Development and Evaluation of a Smart Phone App-based Case Management Model Among ART-naive HIV-infected MSM： A Randomized Controlled Trial
Brief Title: Evaluation of a Smart Phone App-based Case Management Model Among ART-naive HIV-infected MSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Eighth People's Hospital (Unknown)
Responsible Party: Principal Investigator, Gu Jing, Professor of School of Public Health, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017A020212006
Record Dates: First submitted 2019-02-14; First posted 2019-03-01 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: HIV/AIDS
Keywords: case management; men who have sex with men; mhealth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): participants in this arm receive the APP-based case management service and standard-of-care followup service.
  Interventions: Behavioral: APP-based case management service; Behavioral: Standard-of-care followup service
- control group (Active Comparator): participants in the control arm receive standard-of-care followup service
  Interventions: Behavioral: Standard-of-care followup service

INTERVENTIONS:
Behavioral: APP-based case management service — The intervention consists of 4 parts, educational articles, online communication with case managers, supportive service information and visit reminder. Educational articles are both delivered automatically and retrieved by participants. Online communication can also be initiated by participants and case managers. Case managers are request to respond to questions from participants as well as care about medication taking behaviors of each patients during the first month. Supportive service information, which include time, location and charges of service providers will be retrieved by participants, with reminders of available service information scheduled at the beginning of every month. Visit reminders are scheduled at one week before due date.
  Arms: Intervention group
Behavioral: Standard-of-care followup service — When participants initiate HIV antiretroviral treatment (ART), they receive 20-minute ART-related education from the case managers, and have physical examination including blood test, CD4 count, hepatic and renal function tests. Subsequent visits are scheduled at month 1, 2, 3, 6 and 12. During each visit, pills enough to cover days until the next visit will be distributed. And patients will be asked about their medication adherence, high risk behavior and side effects experienced. Any relevant questions from patients will be answered. Physical tests are also included in the routine of each visits.

SUMMARY:
This is a randomized controlled trial about an app-based case management intervention. The intervention is a comprehensive case management approach consisting of the following aspects: articles delivery, online communication with case managers, supportive service information and hospital visits reminders. The aim of this study is to evaluate the efficacy of the intervention among HIV-positive men who have sex with men compared to standard-of-care service.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) are one of the key populations in HIV epidemic. They are characterized by multiple risky sexual behaviors: unprotected anal/oral sex, commercial sex, sex during drug use and multiple partners sexual behavior. In the conservative context of Chinese culture, MSM face a wide variety of psychosocial barriers including: stigma, poor mental health and lack of social support. HIV-positive MSM, not only do they have to deal with external stress about their sexual preference, but they also face the pressure to hide their infection status to avoid discrimination. The aforementioned factors limit their adherence to antiretroviral treatment (ART), and lead to suboptimal treatment outcome. Besides, due to the ART scale-up strategy in China, the existing health system is burdened with increasing numbers of patients, which calls for innovative patient management approach using mobile technology. Moreover, the needs of HIV/AIDS patients are growing complex. So, case management, a comprehensive service model, is adopted to meet the needs of patients with chronic illness, combined with smart phone application (APP) to improve adherence of HIV-positive Chinese men who have sex with men.

This study aims to evaluate the efficacy of an APP-based case management approach on ART adherence. 600 participants will be recruited and randomized into intervention group or control group. The app is called "Trusted Doctor". It allows communication between doctor and patient as well as online patient management including: sharing disease related knowledge, scheduling follow up questionnaire to collect patients' information, visits reminder, free phone calls with phone numbers encrypted. In this study, doctors download the APP, and participants in the intervention group will use Wechat to follow the platform which is connected to Trusted Doctor. Inc server and receive intervention. Wechat is a popular social media that not only allows instant messaging between users, but also provides individuals or groups the function of delivering articles or messages on their own Wechat platform to subscribers. By establishing a unique Wechat platform and link it with the APP, service and relative information can be provided on the daily communication tool. After being screened and informed consent, eligible participants will administer a baseline questionnaire on a tablet and then be randomized into intervention or control group. An identification number will be generated for each participant in this study. Then the intervention group will use Wechat to follow the platform and add contact of case managers. Tutoring about the function of the platform will be provided by investigators. Intervention in this study includes: articles delivery, online communication with case managers, supportive service information and hospital visits reminders. Both the intervention and control group will receive standard-of-care service in the hospital, including medication education after treatment initiation, physical examination and brief counselling scheduled at each hospital visits. Hospital visits are scheduled at month 1/2/3/6/12. Questionnaires are scheduled at baseline, month 1, 3, 6, and 12. Follow-up questionnaires will be delivered through Wechat. The primary outcome is ART adherence and CD4+ T cell count.

ELIGIBILITY:
Inclusion Criteria:

* 1. diagnosed as HIV positive;
* 2. initiate antiretroviral therapy on the day of recruitment;
* 3. was infected through male same-sex behavior;
* 4. has access to internet on a personal mobile phone;
* 5. has a Wechat account and use it daily;
* 6. willing to provide written informed consent;

Exclusion Criteria:

* 1. under severe physical or mental condition which precludes study participation;
* 2. being an inpatient of the hospital;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
self-reported ART medication adherence | month 6 after enrolment
  Measured by visual analogue scale (VAS) ranging from 0 to 100%. The ART medication visual analogue scale is a instrument for patients to rate their dose taken percentages. 100% of doses taken will be regarded as good adherence.
CD4 count | month 6 after enrolment
  measured by flow cytometer during visits to hospitals

SECONDARY OUTCOMES:
Anxiety | baseline and month 1/3/6/12 after enrolment
  Reference： Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Archives of internal medicine 2006; 166(10):1092-1097.
  Anxiety will be measured by Generalized Anxiety Disorder (GAD)-7, including 7 Likert-style items. Response options include "not at all", "several days", "more than half the days", "nearly every day". Scores of 0, 1, 2, and 3 will be assigned to the response categories, respectively. Cronbach's alpha was 0.92. Total score for the scale ranges from 0 to 21. Score will be categorized into 4 level to indicate anxiety level: minimal anxiety (0-4 points), mild anxiety (5-9 points), moderate anxiety (10-14), severe anxiety (15-21)
Depression | baseline and month 1/3/6/12 after enrolment
  Reference: Kroenke K, Spitzer RL. The PHQ-9: A new depression diagnostic and severity measure. Psychiatric Annals 2002; 32(9):509-515.
  The Patient Health Questionnaire (PHQ) -9 is a 9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression. The total of all 9 responses from the PHQ-9 aims to predict the presence and severity of depression. Questions are about the level of interest in doing things, feeling down or depressed, difficulty with sleeping, energy levels, eating habits, self-perception, ability to concentrate, speed of functioning and thoughts of suicide. Responses range from "0" (Not at all) to "3" (nearly every day). A total sum of the responses suggests varying levels of depression. Scores range from 0 to 27. Scores of 10 or higher is suggestive of the presence of depression, with higher score indicating more severe level of depression.
Quality of Life | baseline and month 3/6/12 after enrolment
  Reference: Pedroso B, Gutierrez GL, Duarte E, Pilatti LA, Picinin CT. Quality of life assessment in people living with HIV/AIDS: clarifying the WHOQOL-HIV and WHOQOL-HIV-Bref instruments. In: Global view of HIV infection: InTech; 2011.
  The WHOQOL-HIV BREF is an abbreviated version instrument for evaluation of quality of life specifically designed for people with HIV or AIDS. It contains five extra items specific to PLWHA, and in total contains 31 items. Its items are rated on a 5-points Likert scale, and the available responses are 1 (not at all), 2 (a little) 3 (a moderate amount), 4 (very much) and 5 (an extreme amount). The WHOQOL-HIV BREF contains six domains (physical, psychological, independence, social relations, environment, spiritual/religion/person beliefs) and overall quality of life and general health perceptions. After reverse negatively phrased items, domains and facet scores are scaled in a positive direction where higher scores denote higher quality of life.
ART-related perception | baseline and month 1/3/6/12 after enrolment
  Reference: The Life Windows Project Team. The Life Windows Information Motivation Behavioral Skills ART Adherence Questionnaire (LW-IMB-AAQ). 2006. Center for Health, Intervention, and Prevention. University of Connecticut.
  The LW-IMB-AAQ was developed as a measure of barriers to antiretroviral therapy (ART)adherence among HIV+ patients in clinical care, following the constructs identified in the Information--Motivation--Behavioral Skills (IMB) model of adherence
  The Information and Motivation subscale includes 19 and 10 Likert-style items, respectively. Response options include "Strongly Disagree", "Somewhat Disagree", "Neither Agree nor Disagree", "Somewhat Agree", and "Strongly Agree". Cronbach's alpha was 0.59 and 0.75 in a sample of youth living with HIV, respectively. Higher scores indicate greater knowledge and motivation of ART treatment.
  This subscale includes 14 items. Cronbach's alpha was 0.90. Higher scores indicate greater motivation towards adherence.
High risk sexual behavior | baseline and month 1/3/6/12 after enrolment
  measured by self-selected items including "how many male/female regular/casual partners did you engage in sexual intercourse with during the last month?" And "How frequent did you use condoms during sexual intercourses in the last month with your regular/casual partners?"
Retention in ART | month 1/3/6/12 after enrolment
  kept and missed primary care visits record retrieved from hospital document
HIV RNA viral load | baseline and month 12 after enrolment
  measured by polymerase chain reaction(PCR) during visits to hospitals

OTHER OUTCOMES:
utilization of the case-management service in the intervention group | month 1/3/6/12 after enrolment
  Utilization of the APP will be measured using data retrieved from the APP, including numbers of online communicational messages sent, numbers of each articles being read.
uptake of supportive service | month 1/3/6/12 after enrolment
  will be measured by data from collaborative organization to see if participants use supportive service.
intervention adherence of participants in the intervention group | month 1/3/6/12 after enrolment
  will be measured by a single item asking how frequent they read the educational articles.
sexually transmitted infection | month 1/3/6/12 after enrolment
  number of self-reported sexually transmitted infection (STI) in the past 30 days,
sexual orientation disclosure | month 1/3/6/12 after enrolment
  Status of coming out was coded as involuntarily coming out (outing) (3), voluntarily coming out (2), no coming out with thinking (1), and no coming out and no thinking (0).
HIV infection status disclosure | month 1/3/6/12 after enrolment
  Disclosure of HIV testing was assessed by asking, "Does your main sex partner know that you have been HIV tested?" and "Have you told your main sex partner your HIV test results?"

CONTACTS AND LOCATIONS:
Overall Officials: Jing Gu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available from the principal investigator on reasonable request. Due to the highly sensitive nature of the data collected and the characteristics of this often stigmatized population, no client-level data will be shared until the entire cohort is accrued and completed, even that which is de-identified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after data collection is over
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Fan X, Ning K, Liu C, Zhong H, Lau JTF, Hao C, Hao Y, Li J, Li L, Gu J. Uptake of an App-Based Case Management Service for HIV-Positive Men Who Have Sex With Men in China: Process Evaluation Study. J Med Internet Res. 2023 Apr 26;25:e40176. doi: 10.2196/40176. PMID 37099367
- [Derived] Fan X, She R, Liu C, Zhong H, Lau JTF, Hao C, Li J, Hao Y, Li L, Gu J. Evaluation of smartphone APP-based case-management services among antiretroviral treatment-naive HIV-positive men who have sex with men: a randomized controlled trial protocol. BMC Public Health. 2020 Jan 20;20(1):85. doi: 10.1186/s12889-020-8171-5. PMID 31959139